

#### STATISTICAL ANALYSIS PLAN

**Study Title:** A Phase 2, Open-Label, Randomized Study to Evaluate the

Efficacy and Safety of Andecaliximab (GS-5745) Combined with Nivolumab versus Nivolumab Alone in Subjects with Unresectable or Recurrent Gastric or Gastroesophageal

Junction Adenocarcinoma

Name of Test Drug: Andecaliximab (GS-5745)

Study Number: GS-US-296-2013

**Protocol Version (Date):** Amendment 3

**Analysis Type:** Final

**Analysis Plan Version:** 1.0

**Analysis Plan Date:** 06 Dec 2017

Analysis Plan Author(s): PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

# **TABLE OF CONTENTS**

| TA | BLE O | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF T | ABLES | 4 |
| | | IGURES | |
| LIS | | ABBREVIATIONS | |
| 1. | INTR | ODUCTION | 7 |
| | 1.1. | Study Objectives | 7 |
| | 1.2. | Study Design | |
| | 1.3. | Sample Size and Power | 8 |
| 2. | TYPE | E OF PLANNED ANALYSIS | 9 |
| | 2.1. | Interim Analyses | 9 |
| | 2.2. | Primary Analysis | |
| | 2.3. | Follow-up Analysis | |
| 3. | GEN | ERAL CONSIDERATIONS FOR DATA ANALYSES | 10 |
| | 3.1. | Analysis Sets | 10 |
| | 5.1. | 3.1.1. Intent-to-Treat Analysis Set | |
| | | 3.1.2. Safety Analysis Set | |
| | | 3.1.3. Per-Protocol Analysis Set | |
| | | 3.1.4. Pharmacokinetic Analysis Set | 11 |
| | | 3.1.5. Immunogenicity Analysis Set | |
| | 3.2. | Subject Grouping | |
| | 3.3. | | |
| | 3.4. | Examination of Subject Subgroups | |
| | 3.5. | Multiple Comparisons | |
| | 3.6. | Missing Data and Outliers | |
| | | 3.6.1. Missing Data | |
| | 3.7. | 3.6.2. Outliers | |
| | 3.7. | Analysis Visit Windows | |
| | 5.0. | 3.8.1. Definition of Study Day | |
| | | 3.8.2. Analysis Visit Windows | |
| | | 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit | - |
| | | Window | 17 |
| | 3.9. | Date of Time Point Response and Progression | 18 |
| 4. | SUBJ | ECT DISPOSITION | 19 |
| | 4.1. | Subject Enrollment and Disposition | 19 |
| | 4.2. | Extent of Study Drug Exposure and Adherence | |
| | | 4.2.1. Duration of Exposure to Study Drug | |
| | | 4.2.2. Adherence to Study Drug | |
| | 4.3. | Protocol Deviations | 21 |
| 5. | BASI | ELINE CHARACTERISTICS | 22 |
| | 5.1. | Demographics | |
| | 5.2. | Other Baseline Characteristics | |
| | 5.3. | Medical History | |
| | <u>.</u> . | 5.3.1. Disease History | |
| | 5.4. | Chemotherapy and Radiotherapy Therapy | 23 |

| 6. | EFFIC | CACY AN | ALYSES | 24 |
|---|---|---|---|---|
| | 6.1. | Primary | Efficacy Endpoint. | 24 |
| | 0.1. | 6.1.1. | Statistical Hypothesis for the Primary Efficacy Endpoint | |
| | | 6.1.2. | Analysis for the Primary Efficacy Endpoint | |
| | 6.2. | Seconda | ry Efficacy Endpoint | |
| | | 6.2.1. | Progression-Free Survival | 20 |
| | | 6.2.2. | Overall Survival | 2′ |
| | | 6.2.3. | Duration of Response | 2 |
| | 6.3. | Explorat CCI | tory Efficacy Endpoints | 28 |
| 7. | SAFF | | LYSES | 29 |
| /. | | | | |
| | 7.1. | | Events and Deaths | |
| | | 7.1.1. | Adverse Event Dictionary | |
| | | 7.1.2. | Adverse Event Severity | |
| | | 7.1.3. | Relationship of Adverse Events to Study Drug | |
| | | 7.1.4.<br>7.1.5. | Serious Adverse Events | |
| | | 7.1.5.<br>7.1.6. | Summaries of Adverse Events and Deaths | |
| | 7.2. | | ory Evaluations | |
| | 1.2. | 7.2.1. | Graded Laboratory Values | |
| | | 7.2.1. | Shifts Relative to the Baseline Value | |
| | 7.3. | | eight and Vital Signs | |
| | 7.4. Concomitant Medications | | | |
| | , | 7.4.1. | Prior Medications | |
| | | 7.4.2. | Concomitant Medications. | |
| | 7.5. | Electroc | ardiogram Results | |
| | | 7.5.1. | Investigator Electrocardiogram Assessment | |
| | 7.6. | Other Sa | afety Measures | |
| | 7.7. | Changes | s From Protocol-Specified Safety Analyses | 3- |
| 8. | PHAR | RMACOKI | INETIC (PK) ANALYSES | 3 |
| | 8.1. | PK Sam | ple Collection | 3: |
| | 8.2. | | al Analysis Methods | |
| 9. | IMMU | JNOGENI | ICITY ANALYSES | 30 |
| | 9.1. | $\Lambda D \Lambda S_{0}$ | umple Collection. | 3, |
| | 9.1. | | al Analysis Methods | |
| 10. | BIOM | | ANALYSES | |
| 11. | REFE | RENCES . | | 3 |
| 12. | SOFT | WARE | | 30 |
| 13. | | | 1 | |
| 14. | APPE | NDIX | | 4 |
| | Apper | ndix 1. | List of Laboratory Tests for Safety Analysis | 4 |
| | | ndix 2. | Schedule of Assessments | |

## LIST OF TABLES

| Table 1. | Analysis Visit Windows for Chemistry, Hematology and Vital Signs | 16 |
|---|---|---|
| Table 2. | Analysis Visit Windows for Urinalysis, Pregnancy Test, ECG, and ECOG | 16 |
| Table 3. | Analysis Visit Windows for Thyroid Function Tests (TSH, T3, free T4) | |
| Table 4. | Analysis Visit Windows for Tumor Assessment | 17 |
| Table 5. | Confirmed Overall Response Derivation. | 25 |
| Table 6. | Biomarkers and Assay Testing Methods | 37 |
| | LIST OF FIGURES | |
| Figure 1 | Study Design | 8 |

#### LIST OF ABBREVIATIONS

AE adverse event

ALT alanine aminotransferase
AST aspartate aminotransferase
BLQ below the limit of quantitation

BMI body mass index

CFR Code of Federal Regulations

CI confidence interval
CK creatine kinase
CRF case report form
CSR clinical study report

CTCAE Common Toxicity Criteria for Adverse Events

DCR Disease Control Rate
DMC data monitoring committee

ECG electrocardiogram
ET early termination
FAS Full Analysis Set

GEJ gastroesophageal junction

Hb hemoglobin HLT high-level term

ICH International Conference on Harmonization (of Technical Requirements for Registration of

Pharmaceuticals for Human Use)

ITT intent to treat
LTT lower-level term
LOQ limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

MMR Mismatch Repair

ORR Objective Response Rate

PP per protocol PT preferred term

Q1, Q3 first quartile, third quartile

QRS electrocardiographic deflection between the beginning of the Q wave and termination of the

S wave representing time for ventricular depolarization

QT electrocardiographic interval between the beginning of the Q wave and termination of the T wave

representing the time for both ventricular depolarization and repolarization to occur

QTc QT interval corrected for heart rate

QTcF QT interval corrected for heart rate using Fridericia's formula

RR electrocardiographic interval representing the time measurement between the R wave of

one heartbeat and the R wave of the preceding heartbeat

SAP statistical analysis plan

StD standard deviation

SI (units) international system of units

SOC system organ class

TEAE treatment-emergent adverse event

TFLs tables, figures, and listings
ULN upper limit of normal
VR ventricular rate

WHO World Health Organization

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the interim analysis and clinical study report (CSR) for Study GS-US-296-2013. This SAP is based on the study protocol Amendment 3 dated 16 June 2017 and the electronic case report form (eCRF). The SAP will be finalized before database finalization. Any changes made after the finalization of the SAP will be documented in the CSR.

#### 1.1. Study Objectives

The primary objective of this study is as follows:

• To evaluate and compare the efficacy of andecaliximab (GS-5745) in combination with nivolumab versus nivolumab alone in subjects with recurrent gastric or gastroesophageal junction (GEJ) adenocarcinoma

The secondary objectives of this study are as follows:

- To characterize and compare safety and tolerability of andecaliximab (GS-5745) in combination with nivolumab versus nivolumab alone in subjects with recurrent gastric or GEJ adenocarcinoma
- To characterize the pharmacokinetics (PK) of andecaliximab (GS-5745) in combination with nivolumab

#### 1.2. Study Design

This is a Phase 2, open-label, randomized study comparing andecaliximab (GS-5745) in combination with nivolumab in recurrent gastric and GEJ adenocarcinoma versus nivolumab alone. Approximately 120 subjects will be randomized to either Treatment Arm A: andecaliximab (GS-5745) + nivolumab or Treatment Arm B: nivolumab alone. The primary analysis will be conducted approximately 6 months after the last subject started treatment, when all subjects would have had disease progression or discontinued from the study.

To evaluate safety of the combination drug, an independent Data Monitoring Committee (DMC) will be charged with overseeing the safety of the study. After the first 20 subjects are treated for 8 weeks, the DMC will review all safety data to evaluate for any unexpected toxicities. If the DMC recommends that the combination demonstrates acceptable tolerability, enrollment and randomization will proceed with continued safety oversight from the DMC. Thereafter, review of safety data will be performed at regular intervals as described in the DMC charter.

#### Randomized study:

#### **Treatment Groups:**

- Arm A: Andecaliximab + Nivolumab
- Arm B: Nivolumab

Figure 1. Study Design



#### Randomization and Stratification:

- 1:1 allocation to andecaliximab (GS-5745) + nivolumab versus nivolumab alone through an interactive web response system (IWRS)
- Fixed-block centralized randomization stratified by:
  - PD-L1 positive (>=1% tumor cell staining) versus PD-L1 negative (<1% tumor cell staining)</p>

## 1.3. Sample Size and Power

Assuming the Objective Response Rate (ORR) for subjects treated with nivolumab alone is 25%, 120 subjects in total are needed to detect an improvement of 20% in ORR for subjects treated with andecaliximab (GS-5745) and nivolumab with approximately 83% power at the one-sided significance level of 10% using a Cochran-Mantel-Haenszel (CMH) test with an assumption of common odds ratio for all strata. The assumption of nivolumab ORR is based on the upper bound of the 95% confidence interval of the estimated ORR in CheckMate-032 Study {Le 2016}.

#### 2. TYPE OF PLANNED ANALYSIS

# 2.1. Interim Analyses

No formal interim efficacy analysis is planned.

An external multidisciplinary Data Monitoring Committee (DMC) will review the progress of the study and perform interim reviews of the safety data in order to protect subject welfare and preserve study integrity. To ensure the best interests of the participants, the DMC will recommend to the sponsor if the nature, frequency, and severity of adverse effects associated with the study treatment warrant the early termination of the study, the continuation of the study, or the continuation of the study with modifications.

The initial review will be conducted after 20 subjects have completed through Week 8. Thereafter, review of safety data will be conducted every 6 months.

The DMC's role and responsibilities and the scope of analysis to be provided to the DMC are in a mutually agreed upon charter, which defines the DMC membership, meeting logistics, and meeting frequency.

# 2.2. Primary Analysis

The primary analysis will occur when the last subject is treated for 6 months or discontinued, whichever is earlier.

## 2.3. Follow-up Analysis

After the primary analysis, additional analyses of efficacy and safety may be performed to provide long-term efficacy (overall survival) and safety follow-up.

#### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (StD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

By-subject listings will be presented for all subjects in the Intent-to-Treat (ITT) Analysis Set and sorted by subject ID number, visit date, and time (if applicable). Data collected on log forms, such as AEs, will be presented in chronological order within the subject. The treatment group to which subjects were randomized will be used in the listings. Age, sex at birth, race, and ethnicity will be included in the listings, as space permits.

## 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. The analysis set will be identified and included as a subtitle of each table, figure, and listing.

For each analysis set, the number and percentage of subjects eligible for inclusion will be summarized by treatment group.

# 3.1.1. Intent-to-Treat Analysis Set

The intent-to-treat (ITT) Analysis Set includes all subjects who were randomized in the study. Subjects will be grouped by the treatment to which they were randomized.

The ITT analysis set will be used for subject baseline and disease characteristics and efficacy analyses.

# 3.1.2. Safety Analysis Set

The Safety Analysis Set includes all subjects who took at least 1 dose of study drug (andecaliximab or nivolumab). Subjects will be grouped by the actual treatment received. It will be used for study drug administration and safety analyses.

#### 3.1.3. Per-Protocol Analysis Set

The per-protocol (PP) analysis set includes subjects in the ITT and excludes those who meet any one of the following criteria:

- No documented diagnosis of histologically confirmed adenocarcinoma of the stomach or GEJ with inoperable, locally advanced or metastatic disease, not amenable to curative therapy
- ECOG > 1 at screening

- Did not receive study treatment
- Subjects who have received only neoadjuvant or adjuvant therapy for gastric adenocarcinoma
- Prior treatment with anti-CTLA-4 agents (ipilimumab), anti-PD-1 or anti-PD-L1 agents (pembrolizumab, nivolumab), anti-PD-L2 agents, anti-MMP agents, or other immunomodulatory therapies

The PP analysis set is the secondary analysis set for selected efficacy analyses.

#### 3.1.4. Pharmacokinetic Analysis Set

The Pharmacokinetic (PK) Analysis Set will include all randomized subjects who took at least 1 dose of andecaliximab and have at least 1 nonmissing post dose concentration value reported by the PK laboratory. It will be used for all PK analyses.

#### 3.1.5. Immunogenicity Analysis Set

The Immunogenicity Analysis Set will include all randomized subjects who took at least 1 dose of andecaliximab and have at least 1 nonmissing postdose antidrug antibody (ADA) status reported. This is the primary analysis set for all immunogenicity analyses.

#### 3.2. Subject Grouping

For analyses based on the ITT Analysis Set, subjects will be grouped according to the treatment to which they were randomized. For analyses based on the Safety Analysis Set, subjects will be grouped according to the actual treatment received. The actual treatment received will differ from the randomized treatment only when the actual treatment differs from randomized treatment for the entire treatment duration.

For the PK Analysis Set and Immunogenicity Analysis Set, subjects will be grouped according to the actual treatment they received.

#### 3.3. Strata and Covariates

Subjects will be randomly assigned to treatment groups via the interactive voice or web response system (IXRS) in a 1:1 ratio using a stratified randomization schedule. Stratification will be based on the following variables:

• PD-L1 positive (>=1% tumor cell staining) versus PD-L1 negative (<1% tumor cell staining)

If there are discrepancies in stratification factor values between the IXRS and the Covance lab database, the values recorded in the Covance lab database will be used for analyses.

Efficacy endpoints will be evaluated using stratification factors as covariates or stratification variables for analyses, as specified in Section 6.

In the situation where there is insufficient information in a stratum (ie, if there are < 6 subjects or there is no informative event in a stratum by combined treatment arms), the stratification by PD-L1 will not be applied.

# 3.4. Examination of Subject Subgroups

Primary (ORR) and key secondary (PFS and OS) efficacy endpoints will be examined in the following subgroups if there is sufficient sample size in the subgroup:

| • | Stratification factor PD-L1 status |
|---|---|
| | — <1% tumor cell staining |
| | — >=1% tumor cell staining |
| • | Overall cell PD-L1 staining at baseline |
| | — <1% overall cell PD-L1 staining |
| | — >=1% overall cell PD-L1 staining |
| • | MMR status at baseline |
| | <ul> <li>MMR deficient (Subjects with one or more positive in MSH2, MSH6, MLH1, and PMS2 mutation tests are considered MMR deficient.)</li> </ul> |
| | <ul> <li>MMR proficient (Subjects with all negative in MSH2, MSH6, MLH1, and PMS2 mutation tests are considered MMR proficient.)</li> </ul> |
| • | Primary Site of Tumor |
| | — Gastric |
| | — GEJ |
| • | Number of Prior Anticancer Therapies |
| | <u> </u> |
| | <u> </u> |
| | — 3 |
| | — 4 and above |

- Histological Type
  - Diffuse
  - Other
- Age group
  - \_\_<65
  - **---** >= 65
- Gender
  - Male
  - Female
- Race
  - White
  - Non-White

Adverse events and lab abnormalities will be examined in the following subgroups:

- Age group
  - \_\_<65
  - **---** >= 65
- Gender
  - Male
  - Female
- Race
  - White
  - Non-White

In the situation where there is no responder in a subgroup, odds ratio of ORR within subgroups will not be estimated.

#### 3.5. Multiple Comparisons

There are no adjustments for multiplicity in this study.

#### 3.6. Missing Data and Outliers

#### 3.6.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified. Exceptions are presented in this document.

For missing last dosing date of study drug, imputation rules are described in Section 4.2.1. The handling of missing or incomplete dates for AE onset is described in Section 7.1.5.2, and for prior and concomitant medications in Section 7.4.

#### **3.6.2. Outliers**

Outliers will not be identified during the data management and data analysis process. All data will be included in the data analysis.

#### 3.7. Data Handling Conventions and Transformations

In general, age (in years) on the date of randomization will be used for analyses and presentation in listings. For screen failures, the date the informed consent was signed will be used for age calculation. If only the birth year is collected on the CRF, "01 July" will be used for the unknown birth day and month for the purpose of age calculation. If only birth year and month are collected, "01" will be used for the unknown birth day.

Non-PK data that are continuous in nature but are less than the lower limit of quantitation (LOQ) or above the upper LOQ will be imputed as follows:

- A value that is 1 unit less than the LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "< x" (where x is considered the LOQ). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used to calculate summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used to calculate summary statistics.
- A value that is 1 unit above the LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "> x" (where x is considered the LOQ). Values with decimal points will follow the same logic as above.
- The LOQ will be used to calculate descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the LOQ).

If methods based on the assumption that the data are normally distributed are not adequate, analyses may be performed on transformed data or nonparametric analysis methods may be used, as appropriate.

Natural logarithm transformation will be used for plasma/blood concentrations. Plasma concentration values that are below the limit of quantitation (BLQ) will be presented as "BLQ" in the concentration data listing. Values that are BLQ will be treated as 0 at predose time points, and one-half the value of the LOQ at postbaseline time points.

The following conventions will be used for the presentation of summary and order statistics:

- If at least 1 subject has a concentration value of BLQ for the time point, the minimum value will be displayed as "BLQ."
- If more than 25% of the subjects have a concentration data value of BLQ for a given time point, the minimum and Q1 values will be displayed as "BLQ."
- If more than 50% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, and median values will be displayed as "BLQ."
- If more than 75% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, median, and Q3 values will be displayed as "BLQ."
- If all subjects have concentration data values of BLQ for a given time point, all order statistics (minimum, Q1, median, Q3, and maximum) will be displayed as "BLQ."

#### 3.8. Analysis Visit Windows

#### 3.8.1. Definition of Study Day

Study day will be calculated from the first dosing date of study drug andecaliximab or nivolumab and derived as follows:

- For post dose study days: Assessment Date First Dosing Date + 1
- For days prior to the first dose: Assessment Date First Dosing Date

Therefore, study day 1 is the day of first dose of study drug administration.

#### 3.8.2. Analysis Visit Windows

Subject visits might not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.

The analysis windows for chemistry, hematology and vital signs are provided in Table 1. The analysis windows for urinalysis, pregnancy test, ECG, and ECOG are provided in Table 2. The analysis windows for Thyroid Function Tests (TSH, T3, free T4) are provided in Table 3. The analysis windows for tumor assessment are provided in Table 4.

Table 1. Analysis Visit Windows for Chemistry, Hematology and Vital Signs

| Analysis Visit | Study Day | Lower Limit (inclusive) | Upper Limit (inclusive) |
|---|---|---|---|
| Baseline 1 | | -28 | 1 (before 1 <sup>st</sup> dose) |
| Week 2 15 | | 1 (after first dose) | 21 |
| Week 4 29 | | 22 | 35 |
| Week 6 43 | | 36 | 49 |
| Week X=8, 10, | 7*x+1 | 7x-6 | 7*x + 7 |
| Safety Follow-up | | max (andecaliximab end date,<br>Nivo end date) + 1 | max(andecaliximab end date + 30 days,<br>Nivo end date + 5 months) |

Table 2. Analysis Visit Windows for Urinalysis, Pregnancy Test, ECG, and ECOG

| Analysis Visit Study Day | | Lower Limit (inclusive) | Upper Limit (inclusive) |
|---|---|---|---|
| Baseline 1 | | -28 | 1 (before 1 <sup>st</sup> dose) |
| Week 4 29 | | 1 (after first dose) | 42 |
| Week 8 57 | | 43 | 70 |
| Week 12 85 | | 71 | 98 |
| Week X=16, 20, | 7*x+1 | 7x-13 | 7*x + 14 |
| Safety Follow-up | | max (andecaliximab end date,<br>Nivo end date) + 1 | max(andecaliximab end date + 30 days,<br>Nivo end date + 5 months) |

Note. For pregnancy test, use results from serum test for screening and results from urine test for post-screening visit.

Table 3. Analysis Visit Windows for Thyroid Function Tests (TSH, T3, free T4)

| Analysis Visit Study Day | | Lower Limit (inclusive) | Upper Limit (inclusive) |
|---|---|---|---|
| Baseline | 1 | -28 | 1 (before 1 <sup>st</sup> dose) |
| Week 8 | 57 | 1 (after first dose) | 84 |
| Week 16 | 113 | 85 | 140 |
| Week 24 | 169 | 141 | 196 |
| Week 32, 40, | 7*x+1 | 7x-27 | 7*x + 28 |
| Safety Follow-up | | max (andecaliximab end date,<br>Nivo end date) + 1 | max (andecaliximab end date + 30 days,<br>Nivo end date + 5 months) |

Week X=32, 40, ...

confirmatory

| Analysis Visit | Nominal Study Day | Lower Limit (inclusive) | Upper Limit (inclusive) |
|---|---|---|---|
| Baseline | -28 | Randomization date - 42 | Randomization date |
| Week 8 | 57 | 1 | 84 |
| Week 8 confirmatory | Day of Week 8 visit + 28 | Day of Week 8 visit + 28 | |
| Week 16 | 113 | 85 | 140 |
| Week 16 confirmatory | Day of Week 16 visit + 28 | Day of Week 16 visit + 28 | |
| Week 24 | 169 | 141 | 196 |
| Week 24 confirmatory | Day of Week 24 visit + 28 | Day of Week 24 visit + 28 | |
| Week X=32, 40, | 7*x+1 | 7x-27 | 7*x + 28 |

Table 4. Analysis Visit Windows for Tumor Assessment

Day of Week 32, 40, ...

visit +28

Note: In the rare cases where the screening assessments are after the randomization date but prior to the first dose of study drug, the assessments will be considered as baseline.

Day of Week 32, 40, ...

visit +28

The analysis visit will be used when data are summarized by visit. Any data relating to unscheduled visits will be assigned to a particular visit or time point.

- An unscheduled visit prior to the first dosing of study drug may be included in the calculation of the baseline value, if applicable.
- Unscheduled visits after the first dose of study drug will be included in determining the maximum postbaseline toxicity grade.

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window.

If multiple valid, nonmissing, **continuous** measurements exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

• In general, the baseline value will be the last nonmissing value on or prior to the first dosing date of study drug, unless specified differently. If multiple measurements occur on the same day, the last nonmissing value prior to the time of first dosing of study drug will be considered as the baseline value. If these multiple measurements occur at the same time or the time is not available, the average of these measurements (for continuous data) will be considered the baseline value.

- For post baseline values:
  - The record closest to the nominal day for that visit will be selected.
  - If there are 2 records that are equidistant from the nominal day, the later record will be selected.
  - If there is more than 1 record on the selected day, the average will be taken, unless otherwise specified.

If multiple valid, nonmissing, **categorical** measurements exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- For baseline, the last available record on or prior to the date of the first dose of study drug will be selected. If there are multiple records with the same time or no time recorded on the same day, the value with the lowest severity will be selected (normal will be selected over abnormal for safety ECG findings).
- For post baseline visits, if there are multiple records with the same time or no time recorded on the same day, the value with the worst severity within the window will be selected (abnormal will be selected over normal for safety ECG findings).

# 3.9. Date of Time Point Response and Progression

For subjects who have imaging examinations on various dates that are nevertheless assigned to the same nominal visit window, the following rules apply for the calculation of the endpoint date:

- The response date will be the last date associated with that particular imaging time point.
- The progression date will be the first date associated with that particular imaging time point.

#### 4. SUBJECT DISPOSITION

## 4.1. Subject Enrollment and Disposition

A summary of subject enrollment will be provided by treatment group for each country, investigator, and overall. The summary will present the number and percentage of subjects enrolled. For each column, the denominator for the percentage calculation will be the total number of subjects analyzed for that column.

A similar enrollment table will be provided by randomization stratum. The denominator for the percentage of subjects in the stratum will be the total number of enrolled subjects. If there are discrepancies in the value used for stratification assignment between the IXRS and the clinical database, the value collected in the clinical database will be used for the summary. A listing of subjects with discrepancies in the value used for stratification assignment between the IXRS and the clinical database at the time of data finalization will be provided.

The randomization schedule used for the study will be provided as an appendix to the CSR.

A summary of subject disposition will be provided by treatment group. This summary will present the number of subjects screened, the number of subjects enrolled, and the number of subjects in each of the categories listed below:

- Safety Analysis Set
- Randomized but never dosed
- Continuing study drug
- Completed study drug
- Did not complete study drug with reasons for discontinuation of study drug
- Continuing in tumor assessment
- Completed tumor assessment
- Discontinued tumor assessment before Disease Progression
- Continuing long-term follow-up
- Completed long-term follow-up
- Did not complete long-term follow-up with reasons for discontinuation of long-term follow-up

For the status of study drug and study completion and reasons for discontinuation, the number and percentage of subjects in each category will be provided. The denominator for the percentage calculation will be the total number of subjects in the ITT Analysis Set corresponding to that column.

The following by-subject listings will be provided by subject identification (ID) number in ascending order to support the above summary tables:

• Reasons for study drug, tumor assessment, and long-term follow-up discontinuation

#### 4.2. Extent of Study Drug Exposure and Adherence

Extent of exposure to study drug will be examined by assessing the total duration of exposure to study drug and the level of adherence to the study drug specified in the protocol by component (andecaliximab/nivolumab).

#### 4.2.1. **Duration of Exposure to Study Drug**

Total duration of exposure to study drug will be defined as last dosing date minus first dosing date plus 14, regardless of any temporary interruptions in study drug administration, and will be expressed in weeks using up to 1 decimal place (e.g., 4.5 weeks). If the last study drug dosing date is missing, the latest date among the study drug end date, clinical visit date, laboratory sample collection date, and vital signs assessment date that occurred during the on-treatment period will be used.

The total duration of exposure to study drug will be summarized using descriptive statistics. Summaries will be provided by treatment group for the Safety Analysis Set.

## 4.2.2. Adherence to Study Drug

The total number of doses administered will be summarized using descriptive statistics.

#### 4.2.2.1. On-Treatment Adherence

The level of on-treatment adherence to the study drug regimen will be determined by the total amount of study drug administered relative to the total amount of study drug expected to be administered during a subject's actual on-treatment period based on the study drug regimen, assuming there is no interruption.

The level of on-treatment adherence will be expressed as a percentage using the following formula:

On-Treatment Adherence (%) = 
$$\left(\frac{\text{Total Amount of Study Drug Administered}}{\text{Study Drug Expected to be Administered on Treatment}}\right) \times 100$$

Descriptive statistics for the level of on-treatment adherence with the number and percentage of subjects belonging to adherence categories (e.g.,  $\{<75\%, \ge 75 \text{ to } <90\%, \ge 90\%\}$ ) will be provided by treatment group for the Safety Analysis Set.

No formal statistical testing is planned.

A by-subject listing of study drug administration will be provided by subject ID number (in ascending order) and visit (in chronological order).

#### 4.3. Protocol Deviations

Subjects who did not meet the eligibility criteria for study entry, but enrolled in the study will be summarized regardless of whether they were exempted by the sponsor or not. The summary will present the number and percentage of subjects who did not meet at least 1 eligibility criterion and the number of subjects who did not meet specific criteria by treatment group based on the ITT Analysis Set. A by-subject listing will be provided for those subjects who did not meet at least 1 eligibility (inclusion or exclusion) criterion. The listing will present the eligibility criterion (or criteria if more than 1 deviation) that subjects did not meet and related comments, if collected.

Protocol deviations occurring after subjects entered the study are documented during routine monitoring. The number and percentage of subjects with important protocol deviations by deviation reason (e.g., nonadherence to study drug, violation of select inclusion/exclusion criteria) will be summarized by treatment group for the ITT Analysis Set. A by-subject listing will be provided for those subjects with important protocol deviation.

#### 5. BASELINE CHARACTERISTICS

### 5.1. Demographics

Subject demographic variables (i.e., age, sex, race, and ethnicity) will be summarized by treatment group and overall using descriptive statistics for age, and using number and percentage of subjects for sex, race, and ethnicity. The summary of demographic data will be provided for the ITT Analysis Set.

A by-subject demographic listing, including the informed consent date, will be provided by subject ID number in ascending order.

#### **5.2.** Other Baseline Characteristics

Other baseline characteristics include body weight (in kg), height (in cm), body mass index (BMI; in kg/m²), ECOG, PD-L1 status, and mismatch repair (MMR) status at screening. These baseline characteristics will be summarized by treatment group and overall using descriptive statistics for continuous variables and using number and percentage of subjects for categorical variables. The summary of baseline characteristics will be provided for the ITT Analysis Set. No formal statistical testing is planned.

A by-subject listing of other baseline characteristics will be provided by subject ID number in ascending order.

#### **5.3.** Medical History

General medical history data will be collected at screening and listed only. General medical history data will not be coded.

A by-subject listing of general medical history will be provided by subject ID number in ascending order.

#### 5.3.1. Disease History

A summary of disease-specific medical history will be provided by treatment and overall for the ITT Analysis Set. No formal statistical testing is planned. Variables to be summarized include:

- Primary Tumor Site
- Histology of gastric cancer
- Disease stage at screening
- Differentiation at screening
- Time since diagnosis (months)

The denominator for the percentage of histology of gastric cancer is the number of subjects with gastric cancer. The denominators for the percentage of other variables are the number of subjects in the ITT analysis set corresponding to that column.

A by-subject listing of disease history and surgical procedures will be provided by subject ID number in ascending order.

#### 5.4. Chemotherapy and Radiotherapy Therapy

Prior (neoadjuvant, adjuvant, and metastatic) chemotherapy and radiotherapy will be summarized using descriptive statistics by treatment arm using ITT analysis set.

A by-subject listing of prior anticancer therapy and radiotherapy will be provided by subject ID number in ascending order. A by-subject listing of post-treatment chemotherapy will be provided by subject ID number and time in ascending order.

A by-subject listing of all radiotherapy will be provided by subject ID number and time in ascending order.

#### 6. EFFICACY ANALYSES

Efficacy analysis will be performed based on the ITT Analysis Set. The investigator assessments will be used for analyses of efficacy endpoints.

#### 6.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is objective response rate (ORR), defined as the proportion of subjects with best overall response of complete response (CR) or partial response (PR) after starting study drug but before starting any new chemotherapy or radiotherapy based on revised RECIST 1.1.

As sensitivity analysis, confirmed ORR, defined as the proportion of subjects with best overall response of confirmed complete response (CR) or confirmed partial response (PR) after starting study drug but before starting any new anti-cancer therapy based on revised RECIST 1.1, will also be analyzed. The confirmatory response is required at least 4-week later after the initial CR/PR for confirmed ORR.

Overall response for each visit is derived in the following process. The rules should be applied by the order listed below.

- Response assessments occurring after new anticancer therapy (including radiation therapy), after missing two previous consecutive tumor scans, or after confirmed PD will not be included for ORR analysis.
- If overall response for the first time point of a visit is an imaging PD, in order to differentiate "pseudo-progression (pseudo-PD)" from "definitive progression", the first imaging PD requires confirmation either by another imaging PD at the confirmatory visit at least 4 weeks apart or by the subsequent clinical PD/ radiation therapy. The first imaging PD will be considered as "confirmed PD" by any of the following:
  - The overall response at the confirmatory visit is also PD;
  - No more tumor assessment is available that is 4 weeks apart;
  - The overall response at the confirmatory visit is non-evaluable (NE) and no more tumor assessments follow the confirmatory visit;
  - First imaging PD is followed by subsequent clinical PD or radiation therapy.

Otherwise, the first imaging PD will be "Pseudo PD".

• Both clinical PD and radiation therapy are considered as PD, and no confirmation is required.

The best overall response for each subject across the time points is derived based on the rank CR > PR > SD > pseudo-PD > PD (including clinical PD, confirmed imaging PD, and radiation therapy) > NE.

For confirmed overall response for each visit, in addition to the rules listed above, the following rules should also be applied.

- If overall response for the first time point of a visit (e.g., Week 8) is CR or PR, a confirmatory visit at least 4 weeks later is required. Overall response for the visit is derived based on overall response at the first time point and overall response at the confirmatory visit.
- If overall response for the first time point of a visit is SD/NE, no confirmatory visit is required and the overall response for the visit is SD/NE correspondingly.

The rule for deriving confirmed overall response at each visit is specified in Table 5. The best confirmed overall response for each subject across the time points is derived based on the rank CR confirmed > PR confirmed > CR not confirmed > PR not confirmed > SD > pseudo-PD > PD (including clinical PD, confirmed imaging PD, and radiation therapy) > NE.

**Table 5.** Confirmed Overall Response Derivation

| Overall response at first visit | Overall response at confirmatory visit | Overall response for the time point | Date of Response |
|---|---|---|---|
| | CR | CR confirmed | First visit |
| CR | Responses other than CR or there is no confirmatory visit | CR not confirmed | First visit |
| | CR/PR | PR confirmed | First visit |
| PR | Responses other than CR/PR or there is no confirmatory visit | PR not confirmed | First visit |
| | PD/ clinical PD/ radiation therapy, or there is no confirmatory visit | PD | First visit |
| PD | NE | PD | First visit |
| | Responses other than PD/clinical PD/<br>radiation therapy/NE | pseudo-PD | First Visit |
| NE | Not required | NE | First visit |
| SD | Not required | SD | First visit |

Note: Response after treatment discontinuation does not need to be confirmed.

# 6.1.1. Statistical Hypothesis for the Primary Efficacy Endpoint

The primary efficacy hypothesis is that there is no difference between Treatment Group (Group T) and Control Group (Group C) in ORR. Using  $R_T$  and  $R_C$  to denote the objective response rate of Treatment Group (Group T) and Control Group (Group C), respectively, the statistical hypotheses to be tested in this study will be:

$$H_0$$
:  $R_T = R_C$ 

 $H_1$ :  $R_T > R_C$  (Group T is superior to Group C in terms of ORR)

#### 6.1.2. Analysis for the Primary Efficacy Endpoint

The ORR endpoint will be tested at a two-sided alpha level of 0.2. The ORR will be presented with corresponding 2-sided 80% and 95% exact confidence intervals (CIs) calculated using the Clopper-Pearson method. Odds ratio will also be presented with corresponding 80% and 95% CIs be calculated using the exact Cochran-Mantel-Haenszel (CMH) Chi-square test stratified by screening PD-L1 status. Subjects who do not have sufficient baseline or on-study tumor assessments to characterize response will be counted as non-responders and included in the denominator only.

In addition, the confirmed ORR, defined as the proportion of subjects with best overall response of confirmed CR/confirmed PR will also be presented as a sensitivity analysis. The same analysis methods as for ORR mentioned above will be applied for confirmed ORR.

The analysis for the ORR and confirmed ORR will be performed based on both the ITT Analysis Set and Per Protocol Analysis Set.

#### 6.2. Secondary Efficacy Endpoint

#### **6.2.1.** Progression-Free Survival

Progression free survival (PFS), defined as the interval from the date of randomization to the earlier of the first definitive PD (as defined in section 6.2.1) or death from any cause. The first definitive PD is defined as the first radiation therapy, the first clinical PD, and the first confirmed imaging PD, whichever comes first. Pseudo-PD will not be considered as definitive PD.

Data will be censored on the date of last adequate tumor assessment for subjects (including assessments with a NE outcome):

- who do not have definitive PD or die before study discontinuation, or
- who start new anticancer therapy prior (radiation therapy excluded) to definitive PD or death, or
- who have  $\geq 2$  consecutive missing tumor assessments before definitive PD or death.

Subjects without any adequate baseline tumor assessment are censored on the randomization date. The adequate baseline tumor assessment is defined as the window from (randomization date -35) to randomization date.

PFS in months will be calculated as (date of event/censoring – date of randomization + 1) / 30.4375.

Survival function of PFS is estimated using Kaplan-Meier method and compared using the log-rank test stratified by PD-L1 status at screening. PFS rates at 1, 2, 3, 6, 9, 12 months, and the median with 95% CIs will be derived using Kaplan-Meier methods by treatment arm. Kaplan-Meier curves will also be provided. In addition, hazard ratio (HR) and corresponding 95% CI will be estimated for PFS using the Cox proportional hazards regression model stratified by PD-L1 status at screening.

Follow-up time in months for PFS will be summarized as a continuous variable with descriptive statistics.

- For a subject who is censored from PFS and has discontinued from tumor assessment, duration of PFS follow-up = (Date of Censoring randomization date +1)/30.4375
- For subjects with a definitive PFS event and censored subject with ongoing tumor assessment, duration of PFS follow-up = (Date of analysis cut-off date randomization date +1)/30.4375

Incomplete or missing dates of initiation of anticancer therapy other than the study treatment are imputed as follows:

- If the day is missing but the month and year are available, then the imputed day will be the last day of the month.
- If day and month are missing but year is available, then the imputed day and month will be 01Jan or the last day of the month for the last adequate disease assessment if they have the same year, whichever is later.

The analysis of PFS will be performed based on both the ITT Analysis Set and Per Protocol Analysis Set.

#### 6.2.2. Overall Survival

Overall survival (OS) is defined as interval from the date of randomization to death from any cause. Subjects alive are censored at the last time the subject was known alive.

The survival function of OS is estimated using Kaplan-Meier method and compared using the log-rank test stratified by PD-L1 status at screening. The median, Q1, Q3 estimate of OS and probability of survival at 3, 6, 12, 18, and 24 months from randomization will be provided along with the corresponding 95% CI. In addition, hazard ratio (HR) and corresponding 95% CI will be estimated using Cox proportional hazard regression method stratified by screening PD-L1 status.

Follow-up time in months for OS will be summarized as a continuous variable with descriptive statistics by treatment arm.

- For subjects who discontinued study due to lost to follow-up or withdraw of consent, duration of OS follow-up = (Date of last follow-up – randomization date +1)/30.4375
- For subjects who died and subjects still alive at the time of analysis, duration of OS followup = Date of analysis cut-off date - randomization date +1

The analysis of OS will be performed based on both the ITT Analysis Set and Per Protocol Analysis Set.

# 6.2.3. Duration of Response

Duration of response (DOR) is defined for subjects in the ITT analysis set who are CR/PR prior to new anti-cancer therapy (including radiation therapy) as the interval from the date of the first objective response achieved to the earlier of the first definitive disease progression or death from any cause. The first definitive disease progression is defined in section 6.2.1. The same censoring rules as for PFS will be applied to DOR.

DOR in months = (date of event/censoring - date of first response [CR or PR] + 1) / 30.4375.

Median DOR and 95% CIs will be estimated using Kaplan-Meier methods by treatment arm. Kaplan-Meier curves will also be provided.

#### 6.3. Exploratory Efficacy Endpoints



#### 7. SAFETY ANALYSES

#### 7.1. Adverse Events and Deaths

#### 7.1.1. Adverse Event Dictionary

Clinical and laboratory adverse events (AEs) will be coded using the current version of MedDRA. System organ class (SOC) and preferred term (PT) will be provided in the AE dataset.

# 7.1.2. Adverse Event Severity

Adverse events are graded by the investigator as Grade 1, 2, 3, 4, or 5 according to toxicity criteria specified in the protocol. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings. The missing category will be listed last in summary presentation.

# 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE CRF to the question of "Related to Study Treatment." Relatedness will always default to the investigator's choice, not that of the medical monitor. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if the AEs met the definitions of SAEs that were specified in the study protocol as determined by the investigator. SAEs captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Drug Safety and Public Health Department before data finalization.

#### 7.1.5. Treatment-Emergent Adverse Events

#### 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as both of the following:

- Any AEs with an onset date on or after the study drug start date and up to 30 days after permanent discontinuation of andecaliximab or 5 months after permanent discontinuation of nivolumab
- Any AEs leading to premature discontinuation of andecaliximab or nivolumab

#### 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent. The event is considered treatment emergent if both of the following 2 criteria are met:

- The AE onset is the same as or after the month and year (or year) of the first dosing date of study drug, and
- The AE onset date is the same as or before the month and year (or year) of the date corresponding to 30 days after the date of the last dose of andecaliximab or 5 months after the date of the last dose of nivolumab

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dosing date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

#### 7.1.6. Summaries of Adverse Events and Deaths

Treatment-emergent AEs will be summarized based on the Safety Analysis Set.

The number and percentage of subjects who experienced at least 1 TEAE will be provided and summarized by SOC, HOC, PT, and treatment group. For other AEs described below, summaries will be provided by SOC, PT, and treatment group:

- All TE treatment-related AEs
- TEAEs of Grade 3 or higher (by maximum severity)
- TE Treatment-related AEs of Grade 3 or higher (by maximum severity)
- All TE SAEs
- All TE treatment-related SAEs
- All TEAEs leading to discontinuation of any study drug
- All TEAEs leading to study treatment interruption or dose interruption
- All TEAEs leading to death

A brief, high-level summary of AEs described above will be provided by treatment group and by the number and percentage of subjects who experienced the above AEs.

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC and HT within each SOC, and then by PT in descending order of total frequency within each SOC. For summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual subject during the study.

In addition to the above summary tables, all TEAEs and TE treatment-related AEs will be summarized by PT only, in descending order of total frequency.

Deaths will be summarized by whether it is considered treatment emergent and the cause of the death (AE, due to PD, or other reasons).

In addition, data listings will be provided for the following:

- All AEs, indicating whether the event is treatment emergent
- AEs with Grade 3 or higher
- SAEs
- AEs leading to death
- All deaths
- AEs leading to discontinuation of study drug
- AEs leading to treatment interruption/dose modification

## 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed using qualitative methods. Shift from baseline to worst post-baseline assessment and Grade 3 or higher lab abnormalities will be summarized for the Safety Analysis Set and will include data collected up to the last dose of andecaliximab plus 30 days for subjects who have permanently discontinued andecaliximab or up to the last dose of nivolumab plus 5 months for subjects who have permanently discontinued nivolumab. Severity grade for lab abnormalities are defined by CTCAE 4.03.

A by-subject listing for laboratory test results will be provided by subject ID number and time point in chronological order for hematology, serum chemistry, urinalysis, coagulation, and thyroid function separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the CTCAE severity grade will be flagged in the data listings, as appropriate.

No formal statistical testing is planned.

#### 7.2.1. Graded Laboratory Values

The Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities CTCAE Version 4.03 will be used to assign toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (i.e., increased, decreased) will be presented separately.

#### 7.2.1.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of andecaliximab plus 30 days or nivolumab plus 5 months for subjects who permanently discontinued study drug, or the last available date in the database snapshot for subjects who were still on treatment at the time of an interim analysis. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent.

#### 7.2.1.2. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by lab test and treatment group; subjects will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

- Graded laboratory abnormalities
- Grade 3 or 4 laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with nonmissing postbaseline values up to 30 days after last dosing date of GS5745 or up to 5 months after last dosing date of nivolumab.

A by-subject listing of treatment-emergent Grade 3 or 4 laboratory abnormalities will be provided by subject ID number and time point in chronological order. This listing will include all test results that were collected throughout the study for the lab test of interest, with all applicable severity grades and abnormal flags displayed.

#### 7.2.2. Shifts Relative to the Baseline Value

Shift tables will be presented by showing change in severity grade from baseline to worst post baseline assessment.

# 7.3. Body Weight and Vital Signs

Descriptive statistics will be provided by treatment group for body weight and vital signs as follows:

- Baseline value
- Values at each postbaseline visit
- Change from baseline at each postbaseline visit

A baseline value will be defined as the last available value collected on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3. No formal statistical testing is planned.

A by-subject listing of vital signs and body weight will be provided by subject ID number and time point in chronological order. Body weight will be included in the vital signs listing, if space permits. If not, they will be provided separately.

#### 7.4. Concomitant Medications

Medications collected during the study will be coded using the current version of the [Gilead-modified] World Health Organization (WHO) Drug dictionary.

#### 7.4.1. Prior Medications

A summary of prior medications will not be provided.

#### 7.4.2. Concomitant Medications

Concomitant medications are defined as medications taken while a subject took study drug. Use of concomitant medications will be summarized by Anatomical Therapeutic Chemical (ATC) drug class Level 2 and preferred name using the number and percentage of subjects for each treatment group. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered alphabetically by ATC medical class and then by preferred term in descending overall frequency within each ATC medical class. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medications with a start date prior to or on the first dosing date of study drug and continued to be taken after the first dosing date, or started after the first dosing date but prior to or on the last dosing date of study drug will be considered concomitant medications. Medications started and stopped on the same day as the first dosing date or the last dosing date of study drug will also be considered concomitant. Medications with a stop date prior

to the date of first dosing date of study drug or a start date after the last dosing date of study drug will be excluded from the concomitant medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the date of first study drug administration will be excluded from the concomitant medication summary. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) after the study drug stop date will be excluded from the concomitant medication summary. Medications with completely missing start and stop dates will be included in the concomitant medication summary, unless otherwise specified. Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

All prior and concomitant medications (other than per-protocol study drugs) will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order.

#### 7.5. Electrocardiogram Results

## 7.5.1. Investigator Electrocardiogram Assessment

A by-subject listing for ECG assessment results will be provided by subject ID number and visit in chronological order.

#### 7.6. Other Safety Measures

No additional safety measures are specified in the protocol.

# 7.7. Changes From Protocol-Specified Safety Analyses

There are no deviations from the protocol-specified safety analyses.

# 8. PHARMACOKINETIC (PK) ANALYSES

## 8.1. PK Sample Collection

PK plasma samples will be collected for Arm A only for andecaliximab PK at  $30(\pm 15)$  min after the end of infusion on Day 1; prior to dosing and  $30(\pm 15)$  min after the end of infusion on Day 1 of Weeks 4, 8, 16, 24, and every 3 months thereafter, at the EOT and EOS visits.

#### 8.2. Statistical Analysis Methods

Individual subject concentration for andecaliximab will be listed and summarized using descriptive statistics by treatment. Summary statistics (n, mean, StD, coefficient of variation [%CV], median, min, max, Q1, and Q3) will be presented for individual subject concentration data by time.

Individual concentration data listings and summaries will include all subjects with concentration data. The sample size for each time point will be based on the number of subjects with non-missing concentration data at that time point. The number of subjects with concentration BLQ will be presented for each time point. For summary statistics, BLQ values will be treated as 0 at predose and one-half of the lower limit of quantitation (LLOQ) for postdose time points.

The following tables will be provided for andecaliximab:

• Individual subject concentration data and summary statistics

The following figures may be provided for andecaliximab by treatment:

- Mean (± StD) concentration data versus time (on linear and semilogarithmic scales)
- Median (Q1, Q3) concentration data versus time (on linear and semilogarithmic scales)
- Individual subject concentration versus time (on linear and semilogarithmic scales)

Individual, mean, and median postdose concentration values that are  $\leq$  LLOQ will not be displayed in the figures and remaining points connected.

The following listing will be provided

• PK sampling details by subject, including procedures, differences in scheduled and actual draw times, and sample age will be provided in listings.

## 9. IMMUNOGENICITY ANALYSES

#### 9.1. ADA Sample Collection

For arm A only serum samples for anti-andecaliximab antibody will be collected prior to dosing on Day 1 of week 1, 4, 8, 16, 24, and every 3 months thereafter, EOT, EOS.

# 9.2. Statistical Analysis Methods

Immunogenicity of andecaliximab will be evaluated based upon the positive ADA rate. The number and percentage of subjects exhibiting positive ADA status, defined as ADA presence in serum confirmed in validated assay and reported by bioanalytical laboratory, will be summarized at each specified time point. The number and percentage of subjects exhibiting positive ADA status at any post-andecaliximab time point will also be summarized.

The time to ADA onset will also be assessed. It is defined as the time interval from the date of first dose of andecaliximab to the date positive ADA status is first achieved. The analyses of time to ADA onset will be based on the subjects in the immunogenicity analysis set who have negative ADA status at baseline and achieve positive ADA status at post baseline. Summary statistics (n, mean, StD, coefficient of variation [%CV], median, min, max, Q1, and Q3) will be presented.

Impact of ADA on andecaliximab PK may be evaluated as appropriate. Individual subject andecaliximab predose concentration data may be summarized using descriptive statistics by ADA status (positive or negative) of the same time point. Summary statistics (n, mean, StD, coefficient of variation [%CV], median, min, max, Q1, and Q3) will be presented by ADA status. The number of subjects with concentration BLQ will be presented for each time point. For summary statistics, BLQ values will be treated as 0 at predose. Individual subject andecaliximab predose concentration data versus ADA results may be plotted (on linear and semilogarithmic scales). PK plasma samples meeting below criteria will be included in this analysis:

- Collected after Week 8 Day 1 or later
- Collected 288 384 hours (12 to 16 days) post most recent dose

A by-subject listing for ADA status at each time point and the titer for subjects with positive ADA status will be provided by subject ID number and time point in chronological order.

# 10. BIOMARKER ANALYSES

The following biomarkers will be evaluated whether they are predictive for treatment efficacy. These analyses are exploratory.



# 11. REFERENCES

Le DT, Bendell JC, Calvo E, Kim JW, Ascierto PA, Sharma P, et al. Safety and activity of nivolumab monotherapy in advanced and metastatic (A/M) gastric or gastroesophageal junction cancer (GC/GEC): Results from the CheckMate-032 study [Abstract 06]. J Clin Oncol (ASCO Annual Meeting Abstracts) 2016.

# 12. SOFTWARE

SAS® Software Version 9.X. SAS Institute Inc., Cary, NC, USA.

nQuery Advisor(R) Version X.0. Statistical Solutions, Cork, Ireland.

# 13. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

#### 14. **APPENDIX**

Appendix 1. Appendix 2. List of Laboratory Tests for Safety Analysis Schedule of Assessments

#### Appendix 1. List of Laboratory Tests for Safety Analysis

| Chemistry | Urinalysis | Hematology | Other |
|---|---|---|---|
| Albumin Alkaline phosphatase ALT AST Bicarbonate BUN Calcium Chloride Creatinine <sup>a</sup> Glucose Lipase Amylase Magnesium Phosphorus Potassium | Color and appearance Specific gravity pH Occult blood Protein Glucose Bilirubin Leukocyte esterase Nitrite Urobilinogen Ketones Microscopic <sup>b</sup> | WBC Hemoglobin Hematocrit Platelet ANC Differential Eosinophils Lymphocytes Monocytes Neutrophils | Serum β-hCG or urine pregnancy test <sup>c</sup> Thyroid Function Tests (TSH, T3, freeT4) <sup>d</sup> |
| Sodium Total bilirubin Direct bilirubin Total protein CEA CA125 | | Coagulation PT/INR aPTT | |

ANC = absolute neutrophil count; ALT = alanine aminotransferase; aPTT = Activated Partial Thromboplastin Time; AST = aspartate aminotransferase; BUN = blood urea nitrogen; CEA=carcinoembryonic antigen; β-hCG = beta-human chorionic gonadotropin; INR = International Normalized Ratio; PT = Prothrombin Time; WBC = white blood cell; CA125 = Carbohydrate Antigen 125; TSH = thyroid stimulating hormone; T3 = triiodothyronine; Free T4 = free thyroxine

- a Estimated creatinine clearance (CL<sub>cr</sub>)/glomerular filtration rate will be calculated based on the Cockroft-Gault formula using actual body weight: CL<sub>cr</sub> (mL/min) = (140 age [years])\* weight (kg) / (serum creatinine [mg/dL]\*72). If the subject is female, multiply the quantity by 0.85.
- b Reflex testing based on other abnormalities.
- c Females of child-bearing potential only. Serum pregnancy will be conducted at Screening. Urine pregnancy will be conducted pre-dose on Day 1, every 4 weeks thereafter, at EOT, and EOS, 30-day, and 5-month Safety Follow-up
- d TSH, T3, and free T4 will be tested by the central laboratory at screening. From Week 8 and beyond, T3 and T4 will be tested reflexively based on abnormal TSH results.

# Appendix 2. Schedule of Assessments

| Period | Screening | Randomization Bandomization Ba | | | | | | | | | | | | | EOT <sup>m</sup> | EOT" Disease Progression | EOS | 30 day Safety<br>Follow-up° | 5-month Safety<br>Follow-Up <sup>p</sup> | Long Term<br>Follow-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 to 50 | | Ω | | | | |
| Week | -4 | Day 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 to 96 | | | | | | |
| Window (day) | -28 | 2 11,7 1 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | | | ±7 | ±7 | ±7 | |
| Informed Consent | Х | | | | | | | | | | | | | | | | | | | |
| Medical and Medication<br>History | X | | | | | | | | | | | | | | | | | | | |
| Physical Examination <sup>b</sup> | X | X | | X | | X | | X | | X | | X | | Xs | X | | X | X | | |
| Vital Signs & Weight | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X | X | | |
| ECOG Performance<br>Status <sup>c</sup> | X | X <sup>c</sup> | | Х | | X | | Х | | X | | X | | X <sup>s</sup> | X | | X | X | | |
| 12-lead ECG | X | X | | X | | X | | X | | X | | X | | X <sup>s</sup> | X | | X | | | |
| Adverse events/<br>Concomitant<br>Medications <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| IWRS Registration | Х | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X | | | |
| Study Drug/ Nivolumab<br>Administration <sup>e</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | | | |
| Hematology | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X | X | X | |
| Chemistry | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X | X | X | |
| Thyroid Function Tests (TSH, T3, free T4) | X | | | | | X | | | | X | | | | $X^{t}$ | X | | X | X | X | |

| Period | Screening | Randomization <sup>a</sup> | Treatment | | | | | | | | | | | | | Disease Progression | EOSn | 30 day Safety<br>Follow-up <sup>o</sup> | 5-month Safety<br>Follow-Up <sup>p</sup> | Long Term<br>Follow-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 to 50 | | | | | | |
| Week | -4 | Day 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 to 96 | | | | | | |
| Window (day) | -28 | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | | | ±7 | ±7 | ±7 | |
| Coagulation | X | | | | | | | | | | | | | | X | | X | | | |
| Urinalysis | X | X | | X | | X | | X | | X | | X | | X <sup>s</sup> | X | | X | X | X | |
| Pregnancy Test <sup>f</sup> | X | X | | X | | X | | X | | X | | X | | Xs | X | | X | X | X | |
| Andecaliximab PK <sup>g</sup> | | X | | X | | X | | | | X | | | | Xr | X | | X | | | |
| Anti-Andecaliximab<br>Antibody <sup>h</sup> | | X | | X | | X | | | | X | | | | X <sup>r</sup> | X | | X | | | |
| Blood Biomarkers <sup>i</sup> | X | X | X | X | | X | | | | X | | | | X <sup>r</sup> | | Xi | $X^{i}$ | | | |
| Oral Sampling | | X | | | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | | | | | |
| CT or MRI & Treatment<br>Response Assessment <sup>k</sup> | X | | | | | X | | | | X | | | | X <sup>t</sup> | | X <sup>q</sup> | X | | | |
| Tumor Biopsy <sup>l</sup> | X <sup>l</sup> | | (Wk 5 through Wk 9) | | | | | | | | | | | | X <sup>l</sup> | | | | | |
| Overall Survival and<br>Other Antitumor Therapy | | | | | | | | | | | | | | | | | | | | X <sup>u</sup> |

a Day 1 visit must occur within 3 days following randomization.

b Complete physical examination (PE) to be performed at Screening, EOT and EOS. A modified PE capturing changes from prior exams will be performed at subsequent visits. Height is required at Screening only.

c ECOG performance status on Day 1 may be waived if has been conducted during screening within 4 days of Day 1.

d Adverse events will be assessed and concomitant medications will be recorded at each clinic visit from Screening up to and including the 30-day Safety Follow-up visit or EOS visit whichever is later.

- e For Arm A: Study drug andecaliximab (800 mg) will be administered via IV infusion every 2 weeks over 30 (± 5) min. Nivolumab (3 mg/kg) will be administered via IV infusion following the completion of andecaliximab every 2 weeks over 60 (± 5) min. For Arm B: Nivolumab alone (3 mg/kg) will be administered via IV infusion every 2 weeks over 60 (± 5) min.
- f If applicable (females of child bearing potential). Serum pregnancy testing will be conducted at Screening. Urine pregnancy testing will be conducted pre-dose on Day 1 and every then every 4 weeks, at EOT, and EOS, 30-day, and 5-month Safety Follow-up.
- g For Arm A only, plasma samples will be collected for andecaliximab PK at 30(± 15) min after the end of infusion on Day 1. For Weeks 4, 8, 16, and 24 and every 3 months thereafter, PK will be collected prior to dosing and 30(± 15) min after the end of infusion. It will also be collected at EOT and EOS.
- h For Arm A only, serum samples for anti-andecaliximab antibody will be collected prior to dosing on Day 1, Week 4, Week 8, Week 16, Week 24, and every 3 months thereafter. EOT and EOS.
- i Blood biomarkers will be collected at screening and prior to dosing on Day 1; Week 2; Week 4; Week 8; Week 16; Week 24 and every 3 months thereafter and at progression or EOS.
  - Tumor evaluation by CT or MRI will be performed during screening and approximately every 8 weeks regardless of visit week or dose interruption. Scan at EOS visit is not necessary if restaging scan is performed within the prior 8 weeks. Treatment response assessment will be per RECIST v1.1. For subjects who stop study treatment in the absence of disease progression (eg. experienced unexpected toxicity) and remain on study for follow-up for progression-free survival, tumor evaluation by CT or MRI should continue approximately every 8 weeks until disease progression or initiation of non-study specific anti-neoplastic therapy in the absence of progression, whichever occurs earlier.
- A pretreatment biopsy is requested if archival tumor sample provided to meet Inclusion Criterion #6 is from before the last line of therapy. An on-treatment biopsy is required between Week 5 and Week 9. A biopsy at disease progression is requested, if medically feasible. The sample should be collected by the last clinic visit on study ie EOS or 30 Day Safety Follow-up visit. All biopsies are requested to be from gastric lesions if possible (non-gastric metastatic lesions ok if no gastric lesions possible). See laboratory manual for biopsy specifications and procedures.
- m End of treatment (EOT) assessments will be completed only by subjects who discontinue all treatment prior to disease progression. These assessments should be completed as soon as possible after the decision is made. Every attempt should be made to keep the subject in the study and continue to perform tumor evaluation by CT or MRI approximately every 8 weeks until disease progression.
- n End of study (EOS) assessments will be completed when a subject meets at least 1 of the criteria for study discontinuation (Protocol Section 3.7).
- o The 30-day safety follow-up visit will be performed following the last dose of andecaliximab.
- The 5-month safety follow-up visit will be performed following the last dose of nivolumab.
- If imaging shows progressive disease (PD), it is at the discretion of the investigator to keep the subject on study treatment or to stop study treatment until imaging is repeated ≥4 weeks later in order to confirm PD (see Protocol section 6.2.9).
- r Starting at Week 24, perform every 12 weeks until EOT/EOS.
- s Starting at Week 24, perform every 4 weeks until EOT/EOS.
- t Starting at Week 24, perform every 8 weeks until EOT/EOS.
- u Perform every 3 months until 5 years.